CLINICAL TRIAL: NCT06131697
Title: Effects Of McKenzie Exercises With And Without Mulligan Mobilization On Pain, Disability And Craniocervical Angle In Text Neck Syndrome.
Brief Title: Effects Of McKenzie Exercises With And Without Mulligan Mobilization In Text Neck Syndrome.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/23/0156
Record Dates: First submitted 2023-11-09; First posted 2023-11-14 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Neck Syndrome; Forward Head Posture
Keywords: Text Neck Syndrome; McKenzie Exercises; Sustained Natural Apophyseal Glide; Neck Pain
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants of both group will be informed about the possible risks and potential benefits but they won't know which group they are placed in. The participants must sign consent forms agreeing to the experiment. Concealment will be done via sealed opaque envelopes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- McKenzie Exercises without Mulligan Mobilization (Experimental): McKenzie Exercises including retraction with neck flexion, extension, lateral flexion and rotation exercises.
  Interventions: Other: McKenzie Exercises without Mulligan Mobilization
- McKenzie Exercises with Mulligan Mobilization (Experimental): McKenzie Exercises including retraction with neck flexion, extension, lateral flexion and rotation exercises and Sustained Natural Apophyseal glide.
  Interventions: Other: McKenzie Exercises with Mulligan Mobilization

INTERVENTIONS:
Other: McKenzie Exercises without Mulligan Mobilization — McKenzie Exercises will be comprised of four exercise programs. Retraction with neck flexion, extension, lateral flexion and rotation exercises. Each exercise will be performed with two sets of 10 reps with 10 secs hold twice a week for the time period of four weeks.
  Arms: McKenzie Exercises without Mulligan Mobilization
Other: McKenzie Exercises with Mulligan Mobilization — McKenzie Exercises will be comprised of four exercise programs. Retraction with neck flexion, extension, lateral flexion and rotation exercises. Each exercise will be performed with two sets of 10 reps with 10 secs hold twice a week for the time period of four weeks.
  Along McKenzie exercises Sustained Natural Apophyseal Glide will be given with the tip of thumb placed at an angle of 45° along the eyeball direction reinforced by another thumb. This exercise will be performed for three sets of six repetitions twice a week for the time period of four weeks.
  Arms: McKenzie Exercises with Mulligan Mobilization

SUMMARY:
This study aims to determine the effect of McKenzie exercises with and without Sustained Natural Apophyseal glide on pain, disability, and craniocervical angle in adults with Text neck syndrome.

DETAILED DESCRIPTION:
Text neck syndrome is a condition that results from the repetitive use of electronic devices, causing the neck to flex forward or down for extended periods. This can lead to symptoms such as neck pain, reduced range of motion, weakened muscles, altered joint position, and postural changes such as forward head posture and rounded shoulders.

In this randomized clinical trial, forty eight participants with text neck syndrome will be randomly assigned to one of the two intervention groups:

Group A :McKenzie Exercises without Mulligan mobilization and Group B:McKenzie Exercises with Mulligan mobilization . Randomization will be performed using a convenient random sampling method via sealed opaque envelopes. Each participant will receive a total of eight treatment sessions over a four-week period. The efficacy of the interventions will be assessed at the beginning (first session), conclusion (eight session). Outcome measures, including pain intensity, disability levels and craniocervical angle will be evaluated using the Numeric Pain Rating Scale (NPRS), Neck Disability Index (NDI) and Image J software, respectively. Data will be analyzed using SPSS software version 26. Normality of data will be assessed using the Kolmogorov Smirnov test. For within-group comparisons, either repeated measures ANOVA or the Friedman test will be used. To compare changes between the groups, the independent t-test or Mann-Whitney U test will be applied, depending on the data distribution. The analysis of these outcome measures will provide valuable insights into the impact of the interventions on participants' symptoms and postural alignment.

ELIGIBILITY:
Inclusion Criteria:

Age (18-35 years) Male and Female CVA <49° Using smart phone for more than 5 hours a day Having history of more than 3 months Score more than 3 on NPRS and more than 10 on NDI Score of SAS> 88

Exclusion Criteria:

Neck surgery Spinal infection or inflammatory disorder Diagnosed cases of disc prolapse, stenosis, herniation, spondylolisthesis and osteoporosis, torticollis, scoliosis.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2023-05-10 (Actual); Primary Completion 2023-12-10 (Estimated); Study Completion 2024-01-10 (Estimated)

PRIMARY OUTCOMES:
Numeric pain rating scale (NPRS) | 4th week
  The NPRS is a subjective pain rating scale using an 11-point scale from 0 to 10, where 0 means 'no pain' and 10 means 'intolerable pain'. Participants select the whole number that best represents their level of pain. The reliability is >0.95 with ICC values 0.86-0.95.
Neck disability index (NDI) | 4th week
  NDI has 10 domains covering pain intensity, personal care, lifting, reading, headaches, concentration, work, driving, sleeping, and recreation. Scores range from 0 to 50, with 50 being the greatest levels of dysfunction. It is a valid and realiable tool with ICC=0.98.
Photogrammetry for Craniocervical angle (image j software) | 4th week
  Craniocervical angle can be measured using the lateral photos exposing C7 and the ear. The participants will maintain the natural head posture through the measurement method of self-balance posture. It is the angle made by the line that connects the seventh cervical spine with the tragus and the horizontal line of the seventh cervical spine in the sitting and standing positions. A CVA of <49° is characterized as FHP. Image J is an image processing and analysis program that can read both image file formats and raw formats. It can display, edit, analyze, process, store, and print images, as well as measure distances and angles. It has been introduced as a reliable assessment tool used to measure cervical angles in several studies on forward head posture with ICC of 0.997.

SECONDARY OUTCOMES:
Smartphone Addiction Scale | 1st day
  This scale is used for the recruitment of participants in the study. It is a scale for smartphone addiction that consisted of 6 factors and 33 items with a six-point Likert scale (1: "strongly disagree" and 6: "strongly agree") based on self-reporting. The six factors were daily-life disturbance, positive anticipation, withdrawal, cyberspace-oriented relationship, overuse, and tolerance. Smartphone addiction was categorized as low if total score of a participant was between 33 and 87, intermediate if it was between 88 and 142 and high if score was between 143 and 198.

CONTACTS AND LOCATIONS:
Overall Officials: Ali Raza, Principal Investigator — Riphah International University; Fizza Khan, Principal Investigator — Riphah International University
Locations (1):
- Shalamar Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No